CLINICAL TRIAL: NCT05923229
Title: Moving Mindfully: A MBSR-Centered Approach to Freezing in Parkinson Disease - Randomized Control Trial
Brief Title: Moving Mindfully for Freezing of Gait
Acronym: MM-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gammon M Earhart, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202304132
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Mindfulness
MeSH Terms: conditions — Parkinson Disease | interventions — Weather; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Walking Therapy (MBWT) (Experimental): Participants will receive the MBWT intervention.
  Interventions: Behavioral: Mindfulness Based Walking Therapy (MBWT)
- Freezing of Gait (FOG) Education (Placebo Comparator): Participants will receive educational materials about FOG and track their usual care.
  Interventions: Other: Freezing of Gait (FOG) Education

INTERVENTIONS:
Behavioral: Mindfulness Based Walking Therapy (MBWT) — MBWT is a modified version of the Mindfulness Based Stress Reduction (MBSR) program that incorporates more walking mediations and is acceptable for people with Parkinson disease and freezing of gait.
  Arms: Mindfulness-Based Walking Therapy (MBWT)
Other: Freezing of Gait (FOG) Education — Participants will receive materials to read weekly about FOG and track their usual care regimens.
  Arms: Freezing of Gait (FOG) Education

SUMMARY:
The investigators will conduct an randomized controlled trial (RCT) among people with Parkinson disease (PD) and freezing of gait (FOG) to evaluate the feasibility of a mindfulness intervention compared to a educational program about FOG. FOG is a severe motor disturbance that prevents people from stepping normally and is associated with anxiety, frustration, sedentary behaviors, poorer quality of life, and falls. Mindfulness-Based Stress Reduction (MBSR) is an evidence-based practice that creates a culture to reduce stress and anxiety by increasing conscious awareness and self-compassion. In this study, the investigators will develop a mindfulness-based walking intervention to address both mental health and mobility challenges that constitute FOG.

DETAILED DESCRIPTION:
Conduct pilot randomized clinical trial to evaluate feasibility and acceptability of the standardized Mindfulness Based Walking Therapy (MBWT) program. Using the standardized MBWT protocol devised during earlier aims of this study, the investigators will randomize 24 people with PD+FOG to MBWT or FOG education (i.e., usual care and FOG education), examining feasibility elements.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by a neurologist with idiopathic Parkinson disease;
* age 50 and older;
* a score on the Hoehn & Yahr (H&Y) scale between I-IV;
* history of freezing of gait;
* able to provide informed consent;
* experience fear or worry in relation to their freezing of gait;
* able to walk independently with or without an assistive device for at least five minutes; and
* stable medication regimen for one month prior to enrollment.

Exclusion Criteria:

* have evidence of dementia (Montreal Cognitive Assessment (MOCA) - Telephone Version < 13) to ensure understanding of materials;
* are under consideration for deep brain stimulation surgery within the next six months; neurologic condition other than PD;
* inability to cooperate with the protocol;
* language, visual, or hearing barriers to participation; or
* history of orthopedic or other medical problems that limit ability to participate safely in the intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gammon Earhart, PhD, Principal Investigator — Washington University School of Medicine; Kerri Rawson, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in May 2023 and concluded in August 2023. Recruitment locations included recruitment flyers at physical therapy and movement disorder clinics, health fairs and events, and support groups.
Pre-assignment Details: We consented people via an online format and conducted phone interview screening prior to in-person evaluations. Participants were excluded after the phone interview if they had significant cognitive impairment (MOCA-Telephone Version <13, noted they were not diagnosed with idiopathic Parkinson disease, or could not walk more than five minutes.
Period: Overall Study
Arm/Group | Mindfulness-Based Walking Therapy (MBWT) | Freezing of Gait (FOG) Education
Started | 12 | 12
Completed | 7 | 11
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Health related | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Walking Therapy (MBWT) | Freezing of Gait (FOG) Education | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years of age] | 69.17 (8.45) | 69.83 (7.33) | 69.50 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
New Freezing of Gait Questionnaire (N-FOG) [Mean (Standard Deviation); unit: units on a scale] — The New Freezing of Gait Questionnaire quantifies severity of freezing of gait with a total range of 0 to 28. Higher scores indicate more severe freezing of gait.
  units on a scale | 18.08 (4.87) | 18.58 (4.81) | 18.33 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment of Sample: Number of Participants Recruited
Description: The investigators will count the number of participants recruited to determine if the feasibility objective of recruitment is met. The investigators benchmark for recruitment is defined as recruiting a target sample of 24 participants to randomize.
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Walking Therapy (MBWT) | Freezing of Gait (FOG) Education
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

2. Primary Outcome: Attendance of Participants: Average Number of Participants at Each Session
Description: The investigators will count the number of enrolled participants who were in attendance at each mindfulness session and report the average percentage of participants that attended each mindfulness session over the course of the study to determine if the feasibility objective of attendance is met. The investigators benchmark for attendance is defined as at least 80% of participants attending each session. The number of sessions was 14, we then counted the number of enrolled participants who attended at each session and then averaged that number across the sessions. The unit of measure represents the average number of participants.
Time Frame: 14 weeks
Population: 7 participants who did not withdraw from the 14 week program and 5 participants who withdrew (1 after session 1, 1 after session 2, 1 after session 4, 1 after session 5, 1 after session 7)
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: sessions
Arm/Group | Mindfulness-Based Walking Therapy (MBWT)
Number analyzed (Participants) | 12
Number analyzed (sessions) | 14
percentage of participants | 88.46 [71.43 to 100]

3. Primary Outcome: Retention of Participants: Number of Participants Who Attended 80% of the Sessions or More
Description: The investigators will count the number of participants who attended 11 or more of the 14 sessions (80% of the sessions). Benchmark: Retention is defined as at least 80% of participants attending 80% of the sessions.
Time Frame: 14 weeks
Population: 12 participants (7 participants who did not withdraw and 5 participant who withdrew)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Walking Therapy (MBWT)
Number analyzed (Participants) | 12
Participants | 6

4. Primary Outcome: Adherence: Average Percentage of Hours Participants Practiced Mindfulness at Home
Description: The investigators will ask participants to track the number of hours spent practicing mindfulness at home to determine if the feasibility objective of adherence is met. The investigators benchmark for adherence is as completing 70% of daily home assignment hours. No homework assignments after class 12 (class 13 was the retreat).
Time Frame: 12 weeks
Population: Only 5 of the 7 participants who did not withdraw and 1 participant who did withdraw submitted tracking forms for 6 or more weeks.
Measure: Mean (Full Range); unit: percentage of home assignment hours
Arm/Group | Mindfulness-Based Walking Therapy (MBWT)
Number analyzed (Participants) | 6
percentage of home assignment hours | 89.54 [53 to 247.90]

ADVERSE EVENTS:
Time Frame: 8 months
Description: Injuries that occurred during class time or during the evaluations were reported.
Arm/Group | Mindfulness-Based Walking Therapy (MBWT) | Freezing of Gait (FOG) Education
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Some participants in the Mindfulness-Based Walking Therapy intervention did not return the weekly tracking forms noting the hours they practiced mindfulness at home.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT05923229/Prot_000.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT05923229/ICF_001.pdf